CLINICAL TRIAL: NCT02878200
Title: Reactive Household-based Self-administered Treatment Against Residual Malaria Transmission: a Cluster Randomized Trial
Brief Title: RHOST-cRCT, Reactive Household-based Self-administered Treatment Against Residual Malaria Transmission
Acronym: RHOST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: Institute of Tropical Medicine, Belgium (Other); University of Sheffield (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SCC1488
Record Dates: First submitted 2016-08-22; First posted 2016-08-25 (Estimated); Last update posted 2020-09-07 (Actual); Status verified 2020-09

CONDITIONS: Malaria
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- reactive treatment (Experimental): Household members; defined as those sharing the same sleeping area, in the intervention villages, will be treated with a full course of dihydroartemisinin-piperaquine (DHAP)
  Interventions: Biological: dihydroartemisinin-piperaquine
- standard care (No Intervention): In control villages, no household treatment will be done

INTERVENTIONS:
Biological: dihydroartemisinin-piperaquine — A treatment course of DHAP consists of three doses taken daily. Treatment doses for household members will be prepared based on measured weight
  Other Names: DHAP
  Arms: reactive treatment

SUMMARY:
Reactive treatment of household contacts of a confirmed malaria case has been shown to reduce infection prevalence since the former as they are at an increased risk of infection. However, implementing this on a programmatic scale poses significant pressure on the health system and may not be sustainable without the active involvement of the recipient community. This study investigates a novel approach to reducing residual malaria transmission that combines the elements of active community involvement in reactive treatment of household contacts of a clinical case reporting at a health facility. The investigators hypothesize that in areas of low transmission (prevalence of infection ≤10%), most asymptomatic carriers are clustered around clinical malaria cases in the same households. Also, targeting individuals sharing a sleeping area with diagnosed malaria case will reduce parasite carriage in the community. This is a cluster-randomized trial where villages in Central and Upper Baddibu, North Bank East Region of The Gambia, are randomized to receive either reactive treatment of household contacts following a confirmed case of malaria or standard care, i.e. treatment of index case only. Formative research into community perception and reaction to self-administered treatment will be used to generate, adapt and evaluate messages that encourage adherence and compliance to treatment. This will be tested in the first year of the implementation, and findings used to develop a final model of messages to be implemented in the second year of the study. The primary outcome is the prevalence of malaria infection, determined by molecular methods, in all age groups at the end of the second intervention year and the incidence of clinical malaria during the transmission season.

DETAILED DESCRIPTION:
Achieving malaria elimination presents a challenge because of important gaps in the knowledge about the strategies and tools needed achieve this. While malaria control measures aim to reduce morbidity and mortality in vulnerable populations, interventions to reduce transmission are designed to interrupt transmission of malaria parasites from humans, especially asymptomatic parasite carriers [1], to mosquitoes.

The importance of asymptomatic infections in transmission has grown with the awareness that the majority of the human reservoir of infection are asymptomatic carriers [2] and these are quite difficult to target [3]. Previous malaria elimination campaigns have applied a strategy of mass drug administration: extensive treatment of entire populations, irrespective of their infection status, in one or multiple rounds [4]. Although transmission was interrupted in some cases, albeit temporarily [5], there is a reluctance to apply this method because the evidence of its impact has been mixed. A Cochrane systematic review of MDAs showed that long term reductions were not possible within the current concept and highlighted the need for studies in low- and moderate-transmission settings and studies that could address potential barriers for community uptake, and contribution to the development of drug resistance [6].

More conservative approaches involving screening for infection with a rapid malaria diagnostic test (RDT) and treating only positive individuals; mass screening and treatment, did not have a significant impact on the malaria incidence [7], largely due to low test's sensitivity that would miss a large proportion of infected individuals with low parasite densities. Implementing reactive screening on a programmatic scale puts significant pressure on the health system [8] and available field-based screening tests lack the required sensitivity for low-density parasitaemia seen with asymptomatic infections [9]. More importantly, understanding the local context and adapting intervention strategies may help improve coverage and participation by recipient communities [10].

This study investigates a novel approach to reducing residual malaria transmission that combines the elements of reactive treatment of household contacts of a clinical case reporting at a health facility with the active involvement of both patients and their households. The approach to implementation will be developed through formative research that identifies the optimum means of community engagement that will result in the best possible compliance and adherence to the treatment in the household.

ELIGIBILITY:
Inclusion Criteria:

* Resident in the study area for at least two weeks
* Informed consent to participate in the trial
* willing to receive DHAP (intervention villages)
* Age ≥6 months and weight ≥5kg*

Exclusion Criteria:

* Pregnancy (first trimester only)†
* Known allergies to DHAP
* Known chronic cardiac disease

Min Age: 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 2236 (Actual)
Dates: Start 2016-11-04 (Actual); Primary Completion 2018-12-18 (Actual); Study Completion 2020-07-16 (Actual)

PRIMARY OUTCOMES:
prevalence of malaria infection | 24 months
  the prevalence of malaria infection (determined by molecular methods) in all age groups at the end of the second intervention year

SECONDARY OUTCOMES:
prevalence of clinical (laboratory confirmed) malaria cases | 3-4 months
  the incidence of clinical (laboratory confirmed) malaria cases as detected through the health system; health facilities and village health worker, in both intervention and control clusters
the prevalence of antimalarial drug resistance molecular markers | 4 months and 16 months
  the prevalence of antimalarial drug resistance molecular markers as determined among malaria infected individuals detected at cross-sectional surveys;
treatment coverage | 4 months and 16 months
  treatment coverage as determined by percentage of household members having received and taken at least 80% of the prescribed dose.

CONTACTS AND LOCATIONS:
Overall Officials: Umberto D'Alessandro, MD, Principal Investigator — Medical Research Council Unit, The Gambia
Locations (1):
- Health Centres in North Bank Region, North Bank Region, The Gambia

REFERENCES:
- [Derived] Okebe J, Dabira E, Jaiteh F, Mohammed N, Bradley J, Drammeh NF, Bah A, Masunaga Y, Achan J, Muela Ribera J, Yeung S, Balen J, Peeters Grietens K, D'Alessandro U. Reactive, self-administered malaria treatment against asymptomatic malaria infection: results of a cluster randomized controlled trial in The Gambia. Malar J. 2021 Jun 7;20(1):253. doi: 10.1186/s12936-021-03761-8. PMID 34098984
- [Derived] Okebe J, Ribera JM, Balen J, Jaiteh F, Masunaga Y, Nwakanma D, Bradley J, Yeung S, Peeters Grietens K, D'Alessandro U. Reactive community-based self-administered treatment against residual malaria transmission: study protocol for a randomized controlled trial. Trials. 2018 Feb 20;19(1):126. doi: 10.1186/s13063-018-2506-x. PMID 29463288